CLINICAL TRIAL: NCT01276223
Title: A Multi-Center, Randomized, Double-Masked Evaluation of Anti-Inflammatory Treatment in Patients With Dry Eye
Brief Title: Evaluation of Anti-Inflammatory Treatment in Dry Eye Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-078
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Dry Eye Disease
Keywords: Dry eye; ocular discomfort
MeSH Terms: conditions — Dry Eye Syndromes | interventions — difluprednate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Durezol (Experimental): Difluprednate 0.05% ophthalmic emulsion, 1 drop to the study eye 2 times a day for 4 weeks, followed by 1 drop to the study eye once daily for 1 week to allow for tapering of the steroid exposure.
  Interventions: Drug: Difluprednate 0.05% ophthalmic emulsion
- Vehicle (Placebo Comparator): Difluprednate vehicle, 1 drop to the study eye 2 times a day for 4 weeks, followed by 1 drop to the study eye once daily for 1 week.
  Interventions: Other: Difluprednate vehicle

INTERVENTIONS:
Drug: Difluprednate 0.05% ophthalmic emulsion — Topical ocular steroid
  Other Names: DUREZOL™
  Arms: Durezol
Other: Difluprednate vehicle — Inactive ingredients used as Run-In and placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study was to determine if difluprednate ophthalmic emulsion is effective in reducing the ocular symptoms of dry eye disease, as measured by a global Visual Analog Scale (VAS) discomfort score.

DETAILED DESCRIPTION:
Following Run-In, patients qualifying for treatment were randomized 1:1 to receive Durezol (experimental group) or Vehicle (control group) for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

Normal subjects:

* No known history of dry eye disease.
* Non-contact lens wearer.
* No current use of artificial tears or any other dry eye treatment.

OR

Dry eye patients:

* At least a 6 month history of dry eye.
* Non-contact lens wearer.
* Uses artificial tears.
* Experiences persistent ocular discomfort.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* The presence of any acute infectious or non-infectious ocular conditions in either eye within 1 month of Visit 1.
* Severe Sjogren's Syndrome.
* Lid function abnormalities.
* Use of steroids, tetracycline, doxycycline, etc., within 30 days of Visit 1.
* History of corneal surgery including refractive surgeries.
* History of glaucoma or ocular hypertension
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center at 1-888-451-3937 for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 25 investigative sites located within the US. Participant flow data is presented for all all subjects exposed to product.
Pre-assignment Details: Of the 722 enrolled, 433 subjects did not qualify for Run-In and were exited without exposure to product. Of the 289 entering Run-In, 78 did not qualify for treatment. The 211 patients qualifying for treatment were randomized 1:1 to receive either Durezol or Vehicle.
Groups:
- Run-In Only: Difluprednate vehicle
- Durezol: Difluprednate vehicle (Run-in), followed by difluprednate 0.05% ophthalmic emulsion (treatment)
- Vehicle: Difluprednate vehicle (Run-In), followed by difluprednate vehicle (treatment)
Period: Overall Study
Arm/Group | Run-In Only | Durezol | Vehicle
Started | 78 | 107 | 104
Completed | 67 | 103 | 101
Not Completed | 11 | 4 | 3
Not completed — Adverse Event | 7 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1
Not completed — Pt Decision Unrelated to Adverse Event | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-In Only | Durezol | Vehicle | Total
Number analyzed (Participants) | 78 | 107 | 104 | 289
Age Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.7) | 54.4 (14.8) | 60.1 (13.8) | 58.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 90 | 85 | 242
  Male | 11 | 17 | 19 | 47
Region of Enrollment [Number; unit: participants]
  United States | 78 | 107 | 104 | 289

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Week 0) in Visual Analog Scale (VAS) Global Ocular Discomfort Score Over 4 Weeks
Description: A Visual Analog Scale (VAS) was used by the subject to assess ocular discomfort, both frequency and severity, at baseline (pre-treatment) and weekly thereafter for 4 additional weeks. Each scale was 100 millimeters (mm) in length. The VAS score was calculated by measuring the length in mm from the start of the line to the intersection point of the vertical mark made by the subject. The Global Ocular Discomfort Score is a composite of the two VAS scores, ranging from 0 (very mildly) to 100 (very severely uncomfortable).
Time Frame: Baseline, up to 4 weeks
Population: All subjects randomized to treatment and receiving at least 1 administration of study medication (ITT). Mixed model repeated measure (MMRM) approach was used to handle missing data during randomized treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Durezol: Difluprednate 0.5% ophthalmic emulsion
- Vehicle: Difluprednate vehicle
Arm/Group | Durezol | Vehicle
Number analyzed (Participants) | 107 | 104
units on a scale
  Baseline (Week 0) | 78.3 (14.4) | 76.8 (13.8)
  Change from Baseline to Week 1 | -1.1 (8.8) | -1.7 (12.4)
  Change from Baseline to Week 2 | -4.4 (10.9) | -4.2 (14.7)
  Change from Baseline to Week 3 | -4.5 (13.4) | -4.8 (16.2)
  Change from Baseline to Week 4 | -6.2 (15.1) | -4.7 (16.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (10 months, 15 days).
Description: The safety population includes all subjects exposed to product. Individual subject adverse events, solicited and unsolicited, were collected from time of first instillation of test article (Run-In) until the subject exited the study.
Groups:
- Run-In: Difluprednate vehicle, all patients
- Durezol: Difluprednate 0.05% ophthalmic emulsion
Arm/Group | Run-In | Durezol | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/289 | 1/107 | 1/104
Other Adverse Events (participants affected / at risk) | 47/289 | 12/107 | 3/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In (N=289) | Durezol (N=107) | Vehicle (N=104)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — Not related
Pneumonia (Infections and infestations) | 0 | 0 | 1 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In (N=289) | Durezol (N=107) | Vehicle (N=104)
Eye pain (Eye disorders) | 29 | 1 | 2
Eye irritation (Eye disorders) | 22 | 1 | 2
Intraocular pressure increased (Investigations) | 1 | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.